CLINICAL TRIAL: NCT01634477
Title: Trends of Morbidity and Mortality Among Thai HIV-infected and HIV-uninfected Patients: a Five-year Prospective Cohort Study
Acronym: TNT-HIV
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: HIV Netherlands Australia Thailand Research Collaboration (Network); Bamrasnaradura Infectious Diseases Institute (Other Government); Chulalongkorn University (Other); Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Other Study IDs: TNT-HIV 003
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2021-07

CONDITIONS: HIV Infection; Healthy
Keywords: morbidity; mortality; HIV-infected patients; prospective cohort study; highly active antiretroviral therapy (HAART); opportunistic infections; Non HIV-related illness; cardiovascular disease (CVD); HIV negative patients; Thai HIV-infected patients
MeSH Terms: conditions — HIV Infections; Opportunistic Infections; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-infected patients group: HIV positive
- HIV-uninfected patients group: HIV negative

SUMMARY:
1. To describe the morbidity and clinical characteristics among HIV-infected patients and HIV-uninfected patients.
2. To identify the risk factors for the complication or morbidity among HIV-infected patients and HIV-uninfected patients.
3. To describe the mortality among HIV-infected patients and HIV-uninfected patients.
4. To identify the risk factors for the cause of death among HIV-infected and HIV-uninfected patients.

DETAILED DESCRIPTION:
The information obtained from this study would be very important in planning future holistic care of HIV-infected patients in our institutes as well as in national policy. Results from the study could be used to develop proper long-term management guidelines for people living with HIV (PLHIV) in Thailand targeted at preventable conditions such as metabolic diseases and certain cancers.

ELIGIBILITY:
Inclusion Criteria:

HIV-infected patients group

* HIV positive
* 30 years of age or older, both male and female
* Thai nationality
* Written research informed consent

HIV-uninfected patients group

* HIV un-infected
* 30 years of age or older, both male and female
* Thai nationality
* Written research informed consent

Exclusion Criteria:

HIV-infected patients group

* Systolic BP ≥ 130 or Diastolic BP ≥ 85mm Hg or on the treatment
* Fasting blood sugar > 126 mg/dl or on the treatment
* Proteinuria
* Creatinine > 1.5 mg/dl
* Recent hospitalization
* Patient who are having mental disease HIV-uninfected patients group
* Systolic BP ≥ 130 or Diastolic BP ≥ 85mm Hg or on the treatment
* Fasting blood sugar > 126 mg/dl or on the treatment
* Proteinuria
* Creatinine > 1.5 mg/dl
* Recent hospitalization
* Patient who are having mental disease

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thai HIV-infected patients with and without ART, and HIV negative patients from the Thai Red Cross AIDS Research Centre and Queen Savang Memorial Hospital Institute during January 2010 - December 2014
Sampling Method: Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2010-01; Primary Completion 2020-10 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
morbidity | 60 months
  development of other diseases
HIV related illness | 60 months
  development of opportunistic infection such as Non-Hodkin's lymphoma, Kaposi's sarcoma
Non HIV-related illness | 60 months
  development of Dyslipidemia, Hypertension, DM, CVD , Cancer, osteopenia, osteoporosis, Renal disease, liver disease
mortality | 60 months
  death
CVD | 60 months
  development of CVD

CONTACTS AND LOCATIONS:
Overall Officials: Praphan Phanuphak, MD, Principal Investigator — The Thai Red Cross AIDS Research Centre
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok, Thailand